CLINICAL TRIAL: NCT04090710
Title: Cytoreductive Stereotactic Hypofractionated Radiotherapy With Combination Ipilimumab/Nivolumab for Metastatic Kidney Cancer
Brief Title: SBRT With Combination Ipilimumab/Nivolumab for Metastatic Kidney Cancer
Acronym: CYTOSHRINK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2019-CYTOSHRINK; CA209-7DR (Other Grant/Funding Number: BMS)
Record Dates: First submitted 2019-09-09; First posted 2019-09-16 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: SBRT; Ipilimumab; Nivolumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ipilimumab; Nivolumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Eligible and consenting, newly diagnosed and histologically confirmed intermediate/poor risk metastatic renal cell carcinoma patients with primary disease in-situ will be randomized in a 2:1 fashion to either induction I/N followed by SBRT prior to the second cycle (experimental arm) versus I/N alone (standard arm). Patients will be stratified based on IMDC criteria (intermediate 1-2 versus poor 3-6).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care I/N alone (Active Comparator): induction ipilimumab 1 mg/kg combined with nivolumab 3 mg/kg (I/N) every 3 weeks for cycles 1-4 followed by maintenance treatment with nivolumab 240mg every 2 weeks or 480mg every 4 weeks until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment.
  Interventions: Drug: Ipilimumab/ Nivolumab
- Standard of Care I/N plus primary disease SBRT (Experimental): induction ipilimumab 1 mg/kg combined with nivolumab 3 mg/kg (I/N) every 3 weeks for one cycle, followed by SBRT to the primary disease in-situ, prior to cycle 2-4 of I/N. Patients randomized to SBRT will undergo radiation planning during the first cycle of I/N to their primary kidney mass, and then the radiation will be delivered between cycles 1 and 2 to a dose of 30-40 Gy in 5 fractions every other day over 1.5 weeks. Approximately one week following completion of SBRT, patients will start cycle 2 of immunotherapy as per standard of care. The total time elapsed between the start of cycle 1 and 2 of I/N should be no more than 6 weeks. After completion of up to four cycles of I/N, patients will proceed to standard of care maintenance treatment with nivolumab 240mg every 2 weeks or 480mg every 4 weeks until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment.
  Interventions: Radiation: SBRT + Ipilimumab/Nivolumab

INTERVENTIONS:
Drug: Ipilimumab/ Nivolumab — induction ipilimumab 1 mg/kg combined with nivolumab 3 mg/kg (I/N) every 3 weeks for cycles 1-4 followed by maintenance treatment with nivolumab 240mg every 2 weeks or 480mg every 4 weeks until disease progression
  Other Names: Yervoy/Opdivo
  Arms: Standard of Care I/N alone
Radiation: SBRT + Ipilimumab/Nivolumab — SBRT to the primary disease in-situ, prior to cycle 2-4 of I/N. Patients randomized to SBRT will undergo radiation planning during the first cycle of I/N to their primary kidney mass, and then the radiation will be delivered between cycles 1 and 2 to a dose of 30-40 Gy in 5 fractions every other day over 1.5 weeks.
  Arms: Standard of Care I/N plus primary disease SBRT

SUMMARY:
This trial will evaluate the addition of cytoreductive stereotactic body radiation therapy (SBRT) to standard of care combination ipilimumab and nivolumab (I/N) versus I/N alone for the treatment of metastatic kidney cancer.

DETAILED DESCRIPTION:
This is a multi-centre, open label, phase II randomized clinical trial evaluating SBRT as upfront cytoreductive therapy to the primary renal mass along with combination I/N therapy in patients with intermediate/poor risk mRCC who are not candidates for cytoreductive nephrectomy. Eligible and consenting, newly diagnosed and histologically confirmed intermediate/poor risk mRCC patients based on IMDC criteria with primary disease in-situ will be randomized in a 2:1 fashion to either induction I/N followed by SBRT prior to the second cycle (experimental arm) versus I/N alone (standard arm). Patients will be stratified based on IMDC criteria (intermediate 1-2 versus poor 3-6).

* Standard Arm: induction ipilimumab 1 mg/kg combined with nivolumab 3 mg/kg (I/N) every 3 weeks for cycles 1-4 followed by maintenance treatment with nivolumab 240mg every 2 weeks or 480mg every 4 weeks until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment.
* Experimental Arm: induction ipilimumab 1 mg/kg combined with nivolumab 3 mg/kg (I/N) every 3 weeks for one cycle, followed by SBRT to the primary disease in-situ, prior to cycle 2-4 of I/N. Patients randomized to SBRT will undergo radiation planning during the first cycle of I/N to their primary kidney mass, and then the radiation will be delivered between cycles 1 and 2 to a dose of 30-40 Gy in 5 fractions every other day over 1.5 weeks. Approximately one week following completion of SBRT, patients will start cycle 2 of I/N as per standard of care. The total time elapsed between the start of cycle 1 and 2 of I/N should be no more than 6 weeks. After completion of up to four cycles of I/N, patients will proceed to standard of care maintenance treatment with nivolumab 240mg every 2 weeks or 480mg every 4 weeks until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment.

During treatment (standard and experimental arm) participants will be assessed for radiation toxicity and the occurrence of adverse events. Following treatment, participants will be assessed at a clinic visit every 3 months, for a period of 1 year. Progression free survival will be assessed by CT scan (chest; abdomen and pelvis), which is performed after the final I/N treatment and every 3 months as per standard of care. Participants will be followed for one additional year, seen at 18 and 24 months to assess survival. The planned sample size is 78 study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven renal cell carcinoma of any histology.
2. Imaging proven metastatic disease based on CT or MRI within 10 weeks of screening.
3. Intermediate/poor risk disease based on IMDC criteria (see Appendix II).
4. Primary kidney lesion amenable to SBRT.
5. Eligible for standard of care delivery of ipilimumab and nivolumab (I/N) according to approved product monograph.

Exclusion Criteria:

1. A maximum primary renal lesion size of 20 cm or greater.
2. Candidate for cytoreductive nephrectomy, unless a patient has refused cytoreductive nephrectomy (in this case, a discussion of cytoreductive nephrectomy and patient refusal must be documented).
3. Treatment with prior systemic therapy in the adjuvant or metastatic setting for renal cell carcinoma.
4. Previous abdominal radiation precluding SBRT.
5. Kanofsky Performance (KPS) score below 60 (see Appendix III).
6. History of auto-immune disorder precluding treatment with ipilimumab or nivolumab.
7. History of ataxia telangiectasia or other radiation sensitivity disorders.
8. Chronic corticosteroid use or other chronic immune suppressive therapy. (Participants are permitted the use of topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Adrenal replacement steroid doses of prednisone ≤ 10 mg daily are permitted).
9. Use of medicinal herbal preparations (not including medical cannabis) unless prescribed by a treating physician.
10. Inability to lie flat for at least 30 minutes without moving.
11. Pregnant or lactating women.
12. Geographic inaccessibility for follow-up.
13. Inability to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  The primary outcome of this study is the hazard ratio for progression-free survival (PFS), defined from the date of randomization until the date of progression (PFS truncated at subsequent systemic therapy) as determined by RECIST 1.1, or death due to any cause, whichever comes first. All attempts will be made to follow-up patients for the primary outcome measure for at least one year, even if a patient stops treatment. Patients who do not have a primary outcome event at the time of analysis will be censored on the last date the patient can be confirmed as alive and progression-free.

SECONDARY OUTCOMES:
Subject safety | Date of randomization until 1year post treatment
  Incidence and attribution of deaths
Overall Survival | 2 years
  • Overall survival, defined from the date of randomization to the date of death due to any cause. Patients with no known death date at the time of analysis will be censored on the last date they are confirmed alive.
Objective response rate | 1 year
  • Objective response rate, which is defined as the proportion of randomized subjects who achieve a best response of complete response (CR) or partial response (PR) using the RECIST 1.1 criteria.
Quality of Life: EORTC QLQ-C30 questionnaire | 1 year
  • Quality of life, which will be evaluated using the EORTC QLQ-C30 questionnaire.
Subject safety | 1 Year
  Number of Adverse Events and Serious Adverse Events using NCI CTCAE v5.0
Ipilimumab/ Nivolumab drug tolerability | From the date of randomization until date of first documented disease progression up to 1 year.
  Ipilimumab/Nivolumab treatment discontinuation rates
Ipilimumab/ Nivolumab drug tolerability | From the date of randomization until date of first documented disease progression, up to 1 year.
  Number of doses of Ipilimumab/Nivolumab combination treatment
Ipilimumab/ Nivolumab drug tolerability | From the date of randomization until date of first documented disease progression, up to 1 year.
  Number of Nivolumab maintenance doses
Ipilimumab/ Nivolumab drug tolerability | From the date of randomization until date of first documented disease progression, up to 1 year.
  Time to treatment discontinuation from the date of randomization

OTHER OUTCOMES:
Exploratory Outcomes: Evaluation of baseline and changes during treatment in blood immune signatures | 1 year
  Changes in blood immune signatures through interrogation of circulating blood biomarkers.
Exploratory Outcomes: Evaluation of baseline and changes during treatment in stool microbiome | 1 year
  Changes in stool microbiome using 16S RNA.
Correlation with blood or stool immune signatures | 1 year
  Tumor tissue analysis using immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Aly-Khan Lalani, MD, Principal Investigator — Juravinski Cancer Centre
Locations (7):
- Peter MacCallum Cancer Centre, Melbourne, Australia
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Centre, London, Ontario
  - The Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre- Odette Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No